CLINICAL TRIAL: NCT00642239
Title: A Double-Blind, Placebo-Controlled, Randomized Clinical Trial of Sodium Glycididazole in Concurrent Radiochemotherapy for the Treatment of Thoracic Esophageal Squamous Carcinoma
Brief Title: A Clinical Trial of a Radiation Sensitizer in Radiochemotherapy for Thoracic Esophageal Squamous Carcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Luye Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Lvhua Wang/Professor, Cancer Hospital of Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMNa-ESO-01-2007
Record Dates: First submitted 2008-03-21; First posted 2008-03-25 (Estimated); Last update posted 2008-05-14 (Estimated); Status verified 2008-05

CONDITIONS: Esophageal Carcinoma
Keywords: Sodium Glycididazole, Radiochemotherapy, Esophageal Carcinoma
MeSH Terms: conditions — Esophageal Neoplasms | interventions — sodium glycididazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): Concurrent radiochemotherapy and placebo
  Interventions: Drug: placebo
- 1 (Experimental): concurrent radiochemotherapy and Sodium Glycididazole
  Interventions: Drug: Sodium Glycididazole

INTERVENTIONS:
Drug: placebo — placebo in 100 mL 0.9% NaCl intravenous drip in 30 minutes,then begin radiotherapy in 60 minutes.duration of treatment is 6 weeks.
  Arms: 2
Drug: Sodium Glycididazole — Sodium Glycididazole 700mg/m2 in 100 mL 0.9% NaCl intravenous drip in 30 minutes,then begin radiotherapy in 60 minutes.duration of treatment is 6 weeks.
  Other Names: CMNa
  Arms: 1

SUMMARY:
This multicentered clinical trial is going to find out the radio-sensitization action of sodium glycididazole in radiochemotherapy for esophageal cancer.

DETAILED DESCRIPTION:
Esophageal cancer is one of the most frequent causes of cancer death in the world. The most common type of esophageal cancer is squamous cell carcinoma (SCC) in China. Although concurrent radiochemotherapy is recommended as the standard treatment for advanced esophageal carcinoma, the local failure still reaches up to 44%-54%.

Sodium Glycididazole(CMNa) is a radiosensitive drug for hypoxic tumor cells. Clinical trials showed that CMNa can improve local control rate and survival rate of esophageal cancer. This study is going to confirm the efficacy and safety of CMNa in concurrent radiochemotherapy of radiotherapy and 5-FU+DDP for esophageal squamous carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* photographically and histologically proven thoracic esophageal squamous carcinoma
* stages 2a-3, and stage 4 with only supraclavicular lymph nodes metastasis defined by AJCC(2002)
* radiochemotherapy indication
* measurable tumor
* adequate hematologic, hepatic and renal function
* Karnofsky performance status ≥70
* age more than 18years and less than 70 years

Exclusion Criteria:

* pregnancy and lactation
* significant neurologic disease
* severe liver and renal malfunction,and Significant medical illness
* previous chemotherapy, radiotherapy or immunotherapy
* esophagus hemorrhage and esophagus perforation features

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
tumour local control rate | 6 weeks

SECONDARY OUTCOMES:
survival rate | one year

CONTACTS AND LOCATIONS:
Overall Officials: Lvhua Wang, Doctor, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science
Locations (4):
- China (4):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Center of Sun Yat-sen University, Guangzhou, Guangdong
  - Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing